CLINICAL TRIAL: NCT05516446
Title: Drug Eluting Balloon Angioplasty in Tunisian Population Versus Everolimus Platinum Chrome Stent
Brief Title: Drug Eluting Balloon Angioplasty Versus Everolimus Platinum Chrome Stent
Acronym: DEBATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: General Administration of Military Health, Tunisia (Network)
Collaborators: B. Braun Medical International Trading Company Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: santemilitaire9
Record Dates: First submitted 2022-08-22; First posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Percutaneous Coronary Intervention (PCI); Coronary Artery Disease (CAD); De Novo Stenosis
Keywords: Risk Assessment; Metals; Coronary Artery Disease; Treatment Outcome; Drug-Eluting Stents; Angioplasty, Balloon, Coronary; Randomized Controlled Trials as Topic; Coronary Restenosis
MeSH Terms: conditions — Coronary Artery Disease; Coronary Restenosis

STUDY DESIGN:
Intervention Model Description: Prospective, single-center, randomized and controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEB for de Novo Lesions (Experimental): 1. Preparation of the lesion by pre-dilation or another technique using a balloon undersized by 0.5 mm compared to the reference diameter of the artery and, if necessary, by a second balloon with a balloon/artery ratio of 0.8-1 inflated to 16-18 atm for best results.
  2. when obtaining a stent-like result and in the absence of a major dissection less than grade C, a flow TIMI less than 3 and a residual stenosis of more than 30%, an angioplasty by a drug eluting balloon will be performed for an inflation of 30 seconds at 8-10 atm.
  3. Otherwise, an angioplasty using a drug eluting stent will be proceeded.
  4. Before removing the intracoronary guide, the operator will evaluate by Quantitative Coronary Arteriography (QCA)
     * The post-procedural TIMI flow.
     * the minimal post-procedural luminal diameter in mm.
  Interventions: Device: DEB for de Novo Lesions
- DES for de Novo Lesions (Active Comparator): 1. The preparation of the lesion and the post dilation will be left to the discretion of the operator.
  2. Angioplasty with Drug eluting balloon after pre dilatation will be performed.
  3. Before removing the intracoronary guide, the operator will evaluate by Quantitative Coronary Arteriography (QCA)
     * The post-procedural TIMI flow.
     * the minimal post-procedural luminal diameter in mm.
  Interventions: Device: DES for de Novo Lesions

INTERVENTIONS:
Device: DEB for de Novo Lesions — The surface of the SeQuent® Please NEO balloon is coated with Paclitaxel at a concentration of 3 μg Paclitaxel per mm² of balloon surface. The matrix composed of Paclitaxel and Iopromide (Paccocath technology) allows homogeneous release of the active ingredient through the vessel surface.
  Other Names: a paclitaxel drug-eluting balloon
  Arms: DEB for de Novo Lesions
Device: DES for de Novo Lesions — The latest generation DES : everolimus-eluting platinum-chromium alloy coronary stent system (Promus Premier, Promus Elite)
  Other Names: everolimus-eluting platinum-chromium alloy coronary stent
  Arms: DES for de Novo Lesions

SUMMARY:
Randomized, open-label, single-center, non-inferiority clinical trial to compare late lumen loss (LLL) at 12 months in Tunisian population undergoing coronary percutaneous intervention between Drug Eluting Balloon treated group and Everolimus platinum chrome stent treated group.

DETAILED DESCRIPTION:
Drug eluting stents (DES) leave a permanent metal implant that interferes with vasomotion, endothelial function and vascular remodeling. the rigid structure and the pharmacological properties of DES could overcome acute complications related to balloon dilation and late complications related to in-stent restenosis. However, they do not restore normal arterial function after the procedure.

Drug eluting balloons (DEB) offer an alternative to the implantation of a durable material. They release a transient antiproliferative drug. They promise potential advantages over DES as:

* an ad integrum restitution of the endothelium and its vasomotor properties.
* a reduction of late thrombosis risk.
* the possibility of grafting on the treated segment.
* avoid the problems of side-branch trapped in the treatment of bifurcations.
* improve the profitability of non-invasive imaging (coroscanner, magnetic resonance imaging) during patient follow-up.

DEB is validated for the treatment of in-stent restenosis, especially focal and on small caliber arteries. The use of DEB in de novo lesions has been the subject of several studies. This therapeutic option should be evaluated in the Tunisian context The aim of this clinical trial is to compare the results of angioplasty by DEB (SEQUENT PLEASE) versus last generation DES: coronary stent system in platinum chromium alloy with everolimus elution (Promus Premier and Promus Elite) The Primary endpoint: late lumen loss at 12 months. The Secondary endpoint: the major cardiovascular event rate (MACE).

ELIGIBILITY:
Inclusion Criteria:

* Patients with silent ischemia, stable angina, unstable angina, or non-Q wave myocardial infarction.
* a de Novo lesion on a never treated native artery.
* A reference artery diameter between 2 mm and 4 mm.

Non-inclusion criteria

* Patients with STEMI in the acute phase or presenting a cardiogenic shock.
* Patients with an allergy or a contraindication to double anti-platelet aggregation.
* Pre-menopausal patients not using regularly an oral contraceptives or breast-feeding .
* Patients with severe comorbidity or with an estimated survival of less than 12 months.
* Dissected lesions or spontaneous dissections other than grade A or B requiring DES angioplasty.
* In-stent restenosis.
* Thrombotic lesions.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2021-08-25 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
late lumen loss (LLL) | Follow-up coronary angiography at 12 months after the percutaneous coronary intervention
  late lumen loss between Drug Eluting Balloon treated group and Drug Eluting Stents treated group evaluated by quantitative coronary analysis

SECONDARY OUTCOMES:
rate of major adverse cardiac events (MACE) | 6 months and 12 months after percutaneous coronary intervention
  Major adverse cardiac event defined as the composite of myocardial infarction, target vessel revascularization and cardiac death

CONTACTS AND LOCATIONS:
Overall Officials: Aymen Noamen, MD, Principal Investigator — military hospital of Tunis , Tunis EL manar University, Faculty of medicine of Tunis; Nadhem Hajlaoui, Pr, Study Director — military hospital of Tunis , Tunis EL manar University, Faculty of medicine of Tunis; Wafa Fehri, Pr, Study Chair — military hospital of Tunis , Tunis EL manar University, Faculty of medicine of Tunis
Locations (1):
- Military hospital of Tunis, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhong PY, Ma Y, Shang YS, Niu Y, Bai N, Wang ZL. Efficacy of Drug-Coated Balloon Approaches for de novo Coronary Artery Diseases: A Bayesian Network Meta-Analysis. Front Cardiovasc Med. 2022 Jun 21;9:899701. doi: 10.3389/fcvm.2022.899701. eCollection 2022. PMID 35800174
- [Derived] Hajlaoui N, Noamen A, Ben Amara A, Raddaoui H, Haggui A, Fehri W. Drug-Eluting-Balloon Angioplasty in Tunisian population versus Everolimus-platinum-chrome-stent for de-novo coronary lesion. Tunis Med. 2022 Decembre;100(12):824-829. PMID 37551532